CLINICAL TRIAL: NCT05542537
Title: Nurturing Healthy Teachers: A Cluster-RCT to Improve the Health, Well-being, and Food Security of Early Care and Education (ECE) Professionals
Brief Title: Nurturing Healthy Teachers
Acronym: NHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Brighter Bites (Unknown); Penn State Better Kid Care (Unknown); University of Texas at Austin (Other); Vitamix Foundation (Unknown)
Responsible Party: Principal Investigator, Shreela V Sharma, Professor, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-22-0276
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Nutrition, Healthy; Mental Health Wellness 1; Diabetes Mellitus Risk; Obesity
Keywords: food insecurity; nutrition; healthy eating; wellness; teachers
MeSH Terms: conditions — Obesity | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BB Produce Distribution + BB Nutrition Education + CHF Weekly Wellness Groups + CHF Web-Based Module (Experimental): BB is Brighter Bites. CHF is Create Healthy Futures.
  Interventions: Behavioral: Brighter Bites (BB) Produce Distribution; Behavioral: Brighter Bites (BB) Nutrition Education; Behavioral: Create Healthy Futures (CHF) Weekly Wellness Groups; Behavioral: Create Healthy Futures (CHF) Web-Based Module
- CHF Web-Based Module (Active Comparator): CHF is Create Healthy Futures.
  Interventions: Behavioral: Create Healthy Futures (CHF) Web-Based Module

INTERVENTIONS:
Behavioral: Brighter Bites (BB) Produce Distribution — For 16 weeks in the school year, teachers in participating program schools will receive distributions of 8-10 different types of produce items.
  Arms: BB Produce Distribution + BB Nutrition Education + CHF Weekly Wellness Groups + CHF Web-Based Module
Behavioral: Brighter Bites (BB) Nutrition Education — Brighter Bites Nutrition Education will consist of recipes, food preparation and storage ideas, and tips and tools to budget and plan meals. Teachers will be trained in a nutrition education curriculum, which will be implemented in the program schools as part of the BB program.
  Arms: BB Produce Distribution + BB Nutrition Education + CHF Weekly Wellness Groups + CHF Web-Based Module
Behavioral: Create Healthy Futures (CHF) Weekly Wellness Groups — Peer-facilitators will lead virtual weekly group discussions. Penn State Better Kid Care will train the wellness facilitators.
  Arms: BB Produce Distribution + BB Nutrition Education + CHF Weekly Wellness Groups + CHF Web-Based Module
Behavioral: Create Healthy Futures (CHF) Web-Based Module — Create Healthy Futures Web-Based Module is self-paced and focuses on the following topics: 1) Introduction, 2) Challenges of the food environment, 3) Nutrition and your health, 4) Food culture reform, and 5) Providers' role in creating healthy futures. The Create Healthy Futures module utilizes several educational methods to increase interactivity and engagement, including video footage of content experts, reflection activities, downloadable handouts, and action planning. Each chapter takes approximately 30-40 minutes to complete. The program is delivered on the Better Kid Care On Demand platform, an asynchronous learning management system that provides professional development training for teachers in all 50 states and 69 countries.

SUMMARY:
The purpose of this trial is to compare the impact of a fruit and vegetable access plus nutrition education intervention to a nutrition education-only control on the health, well-being, and food security of early care and education (ECE) professionals. The intervention, called Nurturing Healthy Teachers, combines strategies from two evidence-based programs - Create Healthy Futures (CHF) and Brighter Bites (BB).

DETAILED DESCRIPTION:
The purpose of this trial is to evaluate the impact of the Nurturing Healthy Teachers program on food insecurity, dietary behaviors, mental health, and cardiometabolic health among early care and education (ECE) professionals who teach Pre-Kindergarten or Kindergarten. Nurturing Healthy Teachers is a novel, comprehensive program that combines strategies from two evidence-based programs - Brighter Bites (implemented by Brighter Bites 501c3 non-profit) and Create Healthy Futures (implemented by Penn State Better Kid Care).

1. Brighter Bites (BB) is a 501c3 non-profit organization that implements an evidence-based coordinated school health program that combines access to fresh produce and nutrition education proven to improve dietary intake among preschool and elementary school teachers, low-income children, and their families. For 16 weeks in the school year, Brighter Bites teachers and families receive a weekly distribution of about 20 lbs (50 servings) of primarily donated fresh vegetables, plus weekly healthy recipe tastings, and nutrition education. The program has proven effectiveness at engaging teachers, parents, increasing healthy dietary behaviors and improving the school and home nutrition environment of low-income elementary school children in the short-term.
2. Developed and implemented by Penn State Extension Better Kid Care (BKC), Create Healthy Futures (CHF) is a web-based nutrition education program that targets nutrition knowledge, self-efficacy, mindfulness, and social support to create healthy habits among teachers. CHF also includes facilitated group meetings to reinforce information from the online modules.

The trial will be conducted in 30 elementary schools that have pre-Kindergarten and Kindergarten classes that serve predominantly low-income families in Houston. Schools in the intervention arm (n=15) will receive Brighter Bites plus the complete Create Healthy Futures program including online modules and in-person meetings, and they will be drawn from schools that are already scheduled to receive Brighter Bites during the 2022-2023 school year. Schools in the control arm (n=15) will only receive passive access to the online modules of the Create Healthy Futures program, and they will be drawn from remaining schools across the district, as long as they have not participated in Brighter Bites in the previous two years. The intervention and control programs will be implemented over one school year (9months). Brighter Bites non-profit organization and Penn State Better Kid Care will implement the Nurturing Healthy Teachers program, while UTHealth School of Public Health investigators will conduct the evaluation of the program.

ELIGIBILITY:
Inclusion Criteria for Teachers:

* Employed as a pre-K or kindergarten teaching staff at the participating study schools in the 2022-2023 school year.
* Ability to read English at the 4th grade reading level
* Ability to complete study measures

Exclusion Criteria for Teachers:

* Have recently (in the past 6 months) or are currently participating in an exercise or weight loss program

Inclusion Criteria for Schools:

* Have at least 25 eligible early childhood education (ECE) professionals

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Household Food Insecurity as assessed by the U.S. Department of Agriculture self-report food insecurity survey | baseline
  Household Food insecurity will be measured on an electronically administered using the 10-item self-report previously validated U.S. Department of Agriculture food insecurity survey. The survey will measure food insecurity over the past 30 days. The total score is the sum of affirmative responses to the 10 questions, with a total score range of 0-10. Scores indicate the following about extent of food insecurity:
  * score of zero-High food security
  * score of 1-2-Marginal food security
  * score of 3-5-Low food security
  * score of 6-10-Very low food security
Household Food Insecurity as assessed by the U.S. Department of Agriculture self-report food insecurity measure | 4 months
  Household Food insecurity will be measured on an electronically administered using the 10-item self-report previously validated U.S. Department of Agriculture food insecurity survey. The survey will measure food insecurity over the past 30 days. The total score is the sum of affirmative responses to the 10 questions, with a total score range of 0-10. Scores indicate the following about extent of food insecurity:
  * score of zero-High food security
  * score of 1-2-Marginal food security
  * score of 3-5-Low food security
  * score of 6-10-Very low food security
Household Food Insecurity as assessed by the U.S. Department of Agriculture self-report food insecurity measure | 9 months
  Household Food insecurity will be measured on an electronically administered using the 10-item self-report previously validated U.S. Department of Agriculture food insecurity survey. The survey will measure food insecurity over the past 30 days. The total score is the sum of affirmative responses to the 10 questions, with a total score range of 0-10. Scores indicate the following about extent of food insecurity:
  * score of zero-High food security
  * score of 1-2-Marginal food security
  * score of 3-5-Low food security
  * score of 6-10-Very low food security
Household Food Insecurity as assessed by the U.S. Department of Agriculture self-report food insecurity measure | 14 months
  Household Food insecurity will be measured on an electronically administered using the 10-item self-report previously validated U.S. Department of Agriculture food insecurity survey. The survey will measure food insecurity over the past 30 days. The total score is the sum of affirmative responses to the 10 questions, with a total score range of 0-10. Scores indicate the following about extent of food insecurity:
  * score of zero-High food security
  * score of 1-2-Marginal food security
  * score of 3-5-Low food security
  * score of 6-10-Very low food security

SECONDARY OUTCOMES:
Dietary intake as assessed by self-report survey | baseline
  Dietary intake will be self-reported on an electronically administered survey using a food frequency screener. The survey items will measure the frequency of consumption of various foods including fruits, vegetables, whole grains, protein, water, beverages, desserts, processed food, and candy. Data will be reported categorically as the number of times the surveyed foods were consumed.
Dietary intake as assessed by self-report survey | 9 months
  Dietary intake will be self-reported on an electronically administered survey using a food frequency screener. The survey items will measure the frequency of consumption of various foods including fruits, vegetables, whole grains, protein, water, beverages, desserts, processed food, and candy. Data will be reported categorically as the number of times the surveyed foods were consumed.
Anxiety as assessed by the Generalized Anxiety Disorder 7-item (GAD-7) survey | baseline
  The Generalized Anxiety Disorder 7-item (GAD) survey has a total score from 0 to 21, with a higher score indicating greater anxiety.
Anxiety as assessed by the Generalized Anxiety Disorder 7-item (GAD-7) survey | 9 months
  The Generalized Anxiety Disorder 7-item (GAD) survey has a total score from 0 to 21, with a higher score indicating greater anxiety.
Anxiety as assessed by the Generalized Anxiety Disorder 7-item (GAD-7) survey | 14 months
  The Generalized Anxiety Disorder 7-item (GAD) survey has a total score from 0 to 21, with a higher score indicating greater anxiety.
Anxiety impact as assessed by the impact item of the GAD-7 survey | baseline
  For participants who scored 1 or above on the GAD-7, they will be asked how difficult the anxiety-related issues have made it to do work, take care of things at home, or get along with other people. Data will be reported categorically as number of participants who answered: Not difficult at all; Somewhat difficult; Very difficult; Extremely difficult; Prefer not to say.
Anxiety impact as assessed by the impact item of the GAD-7 survey | 9 months
  For participants who scored 1 or above on the GAD-7, they will be asked how difficult the anxiety-related issues have made it to do work, take care of things at home, or get along with other people. Data will be reported categorically as number of participants who answered: Not difficult at all; Somewhat difficult; Very difficult; Extremely difficult; Prefer not to say.
Anxiety impact as assessed by the impact item of the GAD-7 survey | 14 months
  For participants who scored 1 or above on the GAD-7, they will be asked how difficult the anxiety-related issues have made it to do work, take care of things at home, or get along with other people. Data will be reported categorically as number of participants who answered: Not difficult at all; Somewhat difficult; Very difficult; Extremely difficult; Prefer not to say.
Depression as assessed by the Patient Health 9-item Questionnaire (PHQ-9) | baseline
  The Patient Health 9-item Questionnaire (PHQ-9) has a total score of 0 to 27, with a higher score indicating greater depression.
Depression as assessed by the Patient Health 9-item Questionnaire (PHQ-9) | 9 months
  The Patient Health 9-item Questionnaire (PHQ-9) has a total score of 0 to 27, with a higher score indicating greater depression.
Depression as assessed by the Patient Health 9-item Questionnaire (PHQ-9) | 14 months
  The Patient Health 9-item Questionnaire (PHQ-9) has a total score of 0 to 27, with a higher score indicating greater depression.
Depression impact as assessed by the impact item of the PHQ-9 | baseline
  For participants who scored 1 or above on the PHQ-9, they will be asked how difficult the depression-related issues have made it to do work, take care of things at home, or get along with other people. Data will be reported categorically as number of participants who answered: Not difficult at all; Somewhat difficult; Very difficult; Extremely difficult; Prefer not to say.
Depression impact as assessed by the impact item of the PHQ-9 | 9 months
  For participants who scored 1 or above on the PHQ-9, they will be asked how difficult the depression-related issues have made it to do work, take care of things at home, or get along with other people. Data will be reported categorically as number of participants who answered: Not difficult at all; Somewhat difficult; Very difficult; Extremely difficult; Prefer not to say.
Depression impact as assessed by the impact item of the PHQ-9 | 14 months
  For participants who scored 1 or above on the PHQ-9, they will be asked how difficult the depression-related issues have made it to do work, take care of things at home, or get along with other people. Data will be reported categorically as number of participants who answered: Not difficult at all; Somewhat difficult; Very difficult; Extremely difficult; Prefer not to say.
Well-being as assessed by the 5-item World Health Organization Well-Being Index (WHO-5) | baseline
  The 5-item World Health Organization Well-Being Index (WHO-5) has a total score or 0 -25, with a higher score indicating greater well-being.
Well-being as assessed by the 5-item World Health Organization Well-Being Index (WHO-5) | 9 months
  The 5-item World Health Organization Well-Being Index (WHO-5) has a total score or 0 -25, with a higher score indicating greater well-being.
Well-being as assessed by the 5-item World Health Organization Well-Being Index (WHO-5) | 14 months
  The 5-item World Health Organization Well-Being Index (WHO-5) has a total score or 0 -25, with a higher score indicating greater well-being.
General health as assessed by the general health item of the Centers for Disease Control and Prevention (CDC) Health-related quality of life (HRQoL) 4-item questionnaire (CDC HRQoL-4) | baseline
  Only one item on the CDC HRQoL-4 will be asked, and this is the item related to general health. Participants will be asked if they would say that in general that their health is Excellent, Very good, Good, Fair, Poor, or Prefer not to say. Data will be reported categorically as number of participants who answered: Excellent; Very good; Good; Fair; Poor; Prefer not to say.
General health as assessed by the general health item of the Centers for Disease Control and Prevention (CDC) Health-related quality of life (HRQoL) 4-item questionnaire (CDC HRQoL-4) | 9 months
  Only one item on the CDC HRQoL-4 will be asked, and this is the item related to general health. Participants will be asked if they would say that in general that their health is Excellent, Very good, Good, Fair, Poor, or Prefer not to say. Data will be reported categorically as number of participants who answered: Excellent; Very good; Good; Fair; Poor; Prefer not to say.
General health as assessed by the general health item of the Centers for Disease Control and Prevention (CDC) Health-related quality of life (HRQoL) 4-item questionnaire (CDC HRQoL-4) | 14 months
  Only one item on the CDC HRQoL-4 will be asked, and this is the item related to general health. Participants will be asked if they would say that in general that their health is Excellent, Very good, Good, Fair, Poor, or Prefer not to say. Data will be reported categorically as number of participants who answered: Excellent; Very good; Good; Fair; Poor; Prefer not to say.
Glycosylated hemoglobin (HbA1c) level as assessed by blood test | baseline
  Finger stick blood samples will be obtained from teachers in the school, and HbA1c level in the blood sample will be analyzed.
Glycosylated hemoglobin (HbA1c) level as assessed by blood test | 9 months
  Finger stick blood samples will be obtained from teachers in the school, and HbA1c level in the blood sample will be analyzed.
Blood pressure (systolic) as assessed by automated oscillometric device | baseline
  Blood pressure measurements will be taken using an automated oscillometric device.
Blood pressure (systolic) as assessed by automated oscillometric device | 9 months
  Blood pressure measurements will be taken using an automated oscillometric device.
Blood pressure (diastolic) as assessed by automated oscillometric device | baseline
  Blood pressure measurements will be taken using an automated oscillometric device.
Blood pressure (diastolic) as assessed by automated oscillometric device | 9 months
  Blood pressure measurements will be taken using an automated oscillometric device.
Skin carotenoid level as assessed by The Veggie Meter | baseline
  Skin carotenoid level will be assessed by The Veggie Meter, which is a small, portable non-invasive device that can be clipped to the finger briefly to detect skin carotenoid concentrations in ∼15-20 seconds for a single reading.
Skin carotenoid level as assessed by The Veggie Meter | 9 months
  Skin carotenoid level will be assessed by The Veggie Meter, which is a small, portable non-invasive device that can be clipped to the finger briefly to detect skin carotenoid concentrations in ∼15-20 seconds for a single reading.

CONTACTS AND LOCATIONS:
Overall Officials: Shreela V Sharma, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided